CLINICAL TRIAL: NCT00068328
Title: Observational Cohort Study: Chemotherapy Decisions and Outcomes in Women Age 65 or Older With Operable, Newly Diagnosed Breast Cancer
Brief Title: Chemotherapy Decisions and Outcomes in Older Women With Newly Diagnosed Breast Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-369901; CALGB-369901; CDR0000321396 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IA breast cancer; stage IB breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients participate in interviews over 30-45 minutes at baseline, at 6 months, and at 1 and 2 years.
  Patients are followed annually for at least 5 years.
  Interventions: Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying how older women make treatment decisions and how these decisions affect the outcome of treatment may help doctors plan more effective treatments and improve patient quality of life.

PURPOSE: This clinical trial is studying how a patient's treatment preferences and decisions about chemotherapy affect the outcome of treatment in older women with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between preferences and chemotherapy decisions in women age 65 and over with operable, newly diagnosed breast cancer.
* Determine how factors that could be targets for intervention affect the relationship between preferences and chemotherapy decisions in these patients.
* Determine the relationships between preference-based chemotherapy decisions, quality of life, and satisfaction with treatment decisions in these patients.
* Determine the disease-free survival and competing causes of mortality of these patients.
* Determine the types of physician providers who care for older breast cancer survivors after initial cancer treatment is completed and explore how women decide about which physicians to see.
* Measure quality indicators for the survivorship phase of care and evaluate if quality varies by type of physician provider model.
* Determine if long-term patient-reported satisfaction varies as a function of physician model for providing follow-up care post-treatment.
* Determine whether physician-patient communication and coordination of care after treatment ends mediate follow-up quality and outcomes post-treatment.

OUTLINE: This is a cohort study.

Patients participate in interviews over 30-45 minutes at baseline, at 6 months, and at 1 and 2 years.

Patients are followed annually for at least 5 years.

PROJECTED ACCRUAL: A total of 1,296 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the breast

  * Operable disease
  * Invasive and unilateral tumor
  * No more than 20 weeks since diagnosis
  * T1-4 (tumor size ≥ 1 cm), N0, M0 OR
  * T1-4, N1-3, M0
* No prior carcinoma in situ, lobular carcinoma in situ, ductal carcinoma in situ, or invasive breast cancer
* Hormone receptor status:

  * Any estrogen receptor status

PATIENT CHARACTERISTICS:

Age

* 65 and over

Sex

* Female

Other

* No other malignancy except those for which the patient has completed treatment AND is considered to be at less than 30% risk of recurrence
* History of non-melanoma skin cancer allowed
* Sufficient cognitive function to consent to and complete interviews
* English or Spanish speaking

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Women aged 65 years and older diagnosed with adenocarcinoma of the breast.
Sampling Method: Non-Probability Sample
Enrollment: 1706 (Actual)
Dates: Start 2003-08; Primary Completion 2006-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
quality of life | Up to 5 years

SECONDARY OUTCOMES:
disease free survival | Up to 5 years
mortality rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Mandelblatt, MD, MPH, Study Chair — Lombardi Comprehensive Cancer Center
Locations (85):
- United States (85):
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Pismo Beach, California
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Cancer Center of South Florida Foundation, Incorporated, Lake Worth, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Suniti Medical Corporation, Merrillville, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Oncology Center at St. Joseph Hospital, Nashua, New Hampshire
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - Maria Parham Medical Center, Henderson, North Carolina
  - Southeastern Regional Medical Center, Lumberton, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Duke Health Raleigh Hospital, Raleigh, North Carolina
  - Person Memorial Hospital, Roxboro, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Keyserling Cancer Center at Beaufort Memorial Hospital, Beaufort, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Coastal Cancer Center - Myrtle Beach, Myrtle Beach, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Medical Oncology and Hematology Associates of North Virginia - Fairfax, Fairfax, Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Mandelblatt JS, Faul LA, Luta G, Makgoeng SB, Isaacs C, Taylor K, Sheppard VB, Tallarico M, Barry WT, Cohen HJ. Patient and physician decision styles and breast cancer chemotherapy use in older women: Cancer and Leukemia Group B protocol 369901. J Clin Oncol. 2012 Jul 20;30(21):2609-14. doi: 10.1200/JCO.2011.40.2909. Epub 2012 May 21. PMID 22614985
- [Result] Mandelblatt JS, Sheppard VB, Hurria A, Kimmick G, Isaacs C, Taylor KL, Kornblith AB, Noone AM, Luta G, Tallarico M, Barry WT, Hunegs L, Zon R, Naughton M, Winer E, Hudis C, Edge SB, Cohen HJ, Muss H; Cancer Leukemia Group B. Breast cancer adjuvant chemotherapy decisions in older women: the role of patient preference and interactions with physicians. J Clin Oncol. 2010 Jul 1;28(19):3146-53. doi: 10.1200/JCO.2009.24.3295. Epub 2010 Jun 1. PMID 20516438
- [Result] Mandelblatt J, Sheppard V, Hurria A, et al.: Patient preference as a determinant of breast cancer adjuvant chemotherapy use in older women: CALGB #369901. [Abstract] J Clin Oncol 27 (Suppl 15): A-9544, 2009.
- [Result] Kreling B, Figueiredo MI, Sheppard VL, Mandelblatt JS. A qualitative study of factors affecting chemotherapy use in older women with breast cancer: barriers, promoters, and implications for intervention. Psychooncology. 2006 Dec;15(12):1065-76. doi: 10.1002/pon.1042. PMID 16598833
- [Derived] Bluethmann SM, Alfano CM, Clapp JD, Luta G, Small BJ, Hurria A, Cohen HJ, Sugarman S, B Muss H, Isaacs C, Mandelblatt JS. Cognitive function and discontinuation of adjuvant hormonal therapy in older breast cancer survivors: CALGB 369901 (Alliance). Breast Cancer Res Treat. 2017 Oct;165(3):677-686. doi: 10.1007/s10549-017-4353-y. Epub 2017 Jun 26. PMID 28653250
- [Derived] Mandelblatt JS, Cai L, Luta G, Kimmick G, Clapp J, Isaacs C, Pitcher B, Barry W, Winer E, Sugarman S, Hudis C, Muss H, Cohen HJ, Hurria A. Frailty and long-term mortality of older breast cancer patients: CALGB 369901 (Alliance). Breast Cancer Res Treat. 2017 Jul;164(1):107-117. doi: 10.1007/s10549-017-4222-8. Epub 2017 Mar 31. PMID 28364214